CLINICAL TRIAL: NCT03536689
Title: Randomized Controlled Trial of Amniotic Fluid Index Compared Between After Upright and Left Lateral Decubitus Maternal Position Change
Brief Title: Comparison of Amniotic Fluid Index Between Before and After Maternal Position Change in Upright and Left Lateral Decubitus Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: RAJAAFI001
Record Dates: First submitted 2018-05-14; First posted 2018-05-25 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2018-06

CONDITIONS: Pregnancy Related
Keywords: Amniotic fluid index

STUDY DESIGN:
Intervention Model Description: Factorial 2-by-2 open labeled randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upright maternal position change (Experimental): The participant will be measured by ultrasonograhy for amniotic fluid index in supine position before maternal position change, then she will do the upright position for 5 minute. After 5 minute of upright position , she will lie down in supine position and she will be measured by ultrasonograhy for amniotic fluid index after upright position.
  Interventions: Diagnostic Test: Amniotic fluid index
- Left lateral decubitus maternal position change (Experimental): the participant will be measured by ultrasonograhy for amniotic fluid index in supine position before maternal position change, then she will do the left lateral decubitus position for 5 minutes. After 5 minutes of left lateral decubitus position , she will lie down in supine position and she will be measured by ultrasonograhy for amniotic fluid index after left lateral decubitus position.
  Interventions: Diagnostic Test: Amniotic fluid index

INTERVENTIONS:
Diagnostic Test: Amniotic fluid index — Ultrasonography of the amniotic fluid level in each 4 quadrants of uterus then summerize as one value to measure the quantity of amniotic fluid index
  Other Names: AFI

SUMMARY:
Comparison of amniotic fluid index between before and after maternal position change in Upright and left lateral decubitus maternal position

DETAILED DESCRIPTION:
Amniotic fluid has many important roles in fetal development such as the development of the digestive tract and respiratory system. The quantity of amniotic fluid can be measured by ultrasonography, measuring the deepest pocket in 4 quadrants of uterus then summarize as one value known as "amniotic fluid index"(AFI). The AFI has the normal range between 5-25 cm. The low AFI (< 5 cm) is associated with abnormal fetal heart rate, and the abnormal AFI does affect to the treatment during the antepartum and intrapartum phase. However , there is the study shown that when compared to the single deepest pocket (SDP) , AFI could detect the oligohydramnios more which might led to the unnecessary labor induction or operative delivery without the significant change of perinatal outcome. To increase the accuracy of AFI, we theorize that maternal position change might affect the amniotic fluid position which would increase the visual of the amniotic fluid as well.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 20-34 years whose gestational age was confirmed by ultrasonography before 24 weeks of gestation

Exclusion Criteria:

* Pregnant women with multifetal pregnancy
* Pregnant women who have underlying disease
* Pregnant women who have the history of premature rupture of amniotic membrane
* Pregnant women who have amniotic fluid index below 5 cm (oligohydramnios)
* Pregnant women who have amniotic fluid index more than 25 cm (polyhydramnios)
* Pregnant women whose her baby has the fetal anomaly

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Amniotic fluid index change after maternal position change | 15 minutes
  Amniotic fluid index before and after maternal position change

CONTACTS AND LOCATIONS:
Overall Officials: Tirawat Chotkittikul, MD, Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided